CLINICAL TRIAL: NCT03057834
Title: Exploring the Role of Sarcopenia and Functional Impairment on the Non-Surgical Management of Urinary Incontinence in Older Women
Brief Title: The Urinary Incontinence Treatment Study
Acronym: UNITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00038710; R03AG056460 (NIH)
Record Dates: First submitted 2017-02-10; First posted 2017-02-20 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2021-01

CONDITIONS: Urinary Incontinence; Sarcopenia
MeSH Terms: conditions — Urinary Incontinence; Sarcopenia

STUDY DESIGN:
Intervention Model Description: This will be determined based on the score on the SPPB.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functionally impaired (Active Comparator): Women with urinary incontinence and short physical performance battery score of <9
  Interventions: Behavioral: Pelvic floor muscle exercise
- Functionally normal (Placebo Comparator): Women with urinary incontinence and short physical performance battery score of > 10
  Interventions: Behavioral: Pelvic floor muscle exercise

INTERVENTIONS:
Behavioral: Pelvic floor muscle exercise — Standardized pelvic floor muscle exercise regimen

SUMMARY:
Investigators plan a prospective cohort study with an adaptive design based on physical function status. The design will involve tracking the number of women recruited with physical function impairment and those without any functional impairment. Investigators aim to recruit similar numbers of women in each group. If investigators find unequal numbers, they will adapt recruit strategies based on a woman's functional status.

DETAILED DESCRIPTION:
Investigators plan a prospective cohort study with an adaptive design based on physical function status. The design will involve tracking the number of women recruited with physical function impairment and those without any functional impairment. Investigators aim to recruit similar numbers of women in each group. If they find unequal numbers, they will adapt recruit strategies based on a woman's functional status.

Investigators will compare changes in outcome measures within and between groups after 6 and 12 weeks of pelvic floor muscle exercises (PFME). The change in pelvic floor strength/efficiency will be assessed by repeating the pelvic floor PERFECT assessment and will be compared between groups. Changes in UI symptoms, symptom severity, and impact of UI symptoms on quality of life will be determined using standardized measures described above. Data analysis will define associations between changes in PERFECT measures and the change in UI episodes (based on 3-day voiding diary), severity, and type (based on QUID-7), and impact on quality of life (PFIQ-7) within and between groups. Objective measurement of lower-extremity strength will inform the relationship between lower-extremity strength, pelvic floor strength, and UI symptoms at baseline and the 6-week visit.

ELIGIBILITY:
Inclusion Criteria:

* Women, age 70 years or older
* Diagnosis of Urinary Incontinence (defined by the QUID assessment as having subscale score for stress ≥4, and/or urge score ≥ 6)
* Willing and able to be compliant with pelvic floor muscle exercise intervention (standard of care) for 12 weeks and to log compliance
* Willing and able to undergo an extensive physical function evaluation

Exclusion Criteria:

* Prior surgical intervention for urinary incontinence within the past 12 months
* Hysterectomy within 12 months
* Diagnosis of:
* Pelvic Organ Prolapse beyond the hymenal ring
* Urogenital Fistula
* Neurogenic Overactive Bladder (associated with a diagnosis of Multiple -Sclerosis or Stroke within past 12 months)
* Incomplete Bladder Emptying/Urinary Retention with PVR >150 ml (measured by bladder scan)
* Requires assisted device (4 point cane, walker) for ambulation all /most of the time or wheelchair bound
* Having significant cognitive impairment or dementia
* Unsafe to exercise (severe cardiopulmonary disease)
* Unable/unwilling to provide informed consent
* Determined otherwise ineligible by the principal investigator

Min Age: 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Must be born a woman due to the nature of the intervention investigators are studying.
Enrollment: 70 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candace Parker-Autry, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parker-Autry C, Neiberg R, Leng XI, Matthews CA, Dumoulin C, Kuchel G, Kritchevsky SB. Examining the Role of Nonsurgical Therapy in the Treatment of Geriatric Urinary Incontinence. Obstet Gynecol. 2022 Aug 1;140(2):243-251. doi: 10.1097/AOG.0000000000004852. Epub 2022 Jul 6. PMID 35852275

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Functionally Impaired | Functionally Normal
Started | 33 | 37
Week 6 | 28 | 30
Week 12 | 25 | 29
Completed | 8 | 8
Not Completed | 25 | 29
Not completed — Withdrawal by Subject | 25 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Functionally Impaired | Functionally Normal | Total
Number analyzed (Participants) | 33 | 37 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.9 (6.4) | 76 (4.1) | 76.9 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 37 | 70
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 27 | 32 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 37 | 70
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Weight (kg) / Height (m)^2] | 33.6 (14.5) | 27.5 (5.8) | 30.53 (3.05)

OUTCOME MEASURES:

1. Primary Outcome: Number of Urinary Incontinence Episodes
Description: Using a three-day voiding diary
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: number of incontinence episodes
Arm/Group | Functionally Impaired | Functionally Normal
Number analyzed (Participants) | 33 | 37
number of incontinence episodes | 4.3 (0.6) | 2.7 (0.6)

2. Primary Outcome: Number of Urinary Incontinence Episodes
Description: Using a three-day voiding diary
Time Frame: week 6
Measure: Mean (Standard Deviation); unit: number of incontinence episodes
Arm/Group | Functionally Impaired | Functionally Normal
Number analyzed (Participants) | 28 | 30
number of incontinence episodes | 3.4 (0.6) | 2.3 (0.6)

3. Primary Outcome: Number of Urinary Incontinence Episodes
Description: Using a three-day voiding diary
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: number of incontinence episodes
Arm/Group | Functionally Impaired | Functionally Normal
Number analyzed (Participants) | 25 | 29
number of incontinence episodes | 3.5 (0.6) | 2.4 (0.6)

4. Secondary Outcome: Power of Contractions
Description: measurement of strength using perineometer
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Functionally Impaired | Functionally Normal
Number analyzed (Participants) | 25 | 29
cmH2O | 19.3 (13.3) | 29.3 (16)

5. Secondary Outcome: Endurance
Description: measure of how long they can hold contraction
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: time in seconds
Arm/Group | Functionally Impaired | Functionally Normal
Number analyzed (Participants) | 25 | 29
time in seconds | 4.4 (2.0) | 4.7 (1.9)

6. Secondary Outcome: Repetition of Contractions
Description: how many repetitions can they sustain
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: number of repetitions
Arm/Group | Functionally Impaired | Functionally Normal
Number analyzed (Participants) | 25 | 29
number of repetitions | 9.1 (1.9) | 8.8 (1.9)

7. Secondary Outcome: Number of Fast Contractions
Description: number of fast contractions that can be repeated
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: number of fast contractions
Arm/Group | Functionally Impaired | Functionally Normal
Number analyzed (Participants) | 25 | 29
number of fast contractions | 4.3 (1.7) | 4.7 (1.5)

8. Other Pre Specified Outcome: Pelvic Organ Prolapse
Description: measured using the standardized Pelvic Organ Prolapse Quantification (POP-Q) system
Time Frame: baseline, week 12
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Short Physical Performance Battery (expSPPB)--Gait Speed
Description: expSPPB scores range from zero to 12 possible points. SPPB score of 0 indicates the lowest physical performance, and a score of 12 indicates the highest performance
Time Frame: week 12
Reporting Status: Not Posted

10. Other Pre Specified Outcome: 400 Meter Walk
Description: measurement of exercise tolerance
Time Frame: week 12
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Isokinetic Dynamometer
Description: maximal isokinetic knee extensor strength in the right leg will be measured at speeds of 60 degrees/sec. The left leg will be used if there is a reason not to measure the right leg.
Time Frame: week 12
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Postural Sway
Description: Center-of-Pressure (COP) trajectory data will be collected using an Advanced Mechanical Incorporated (AMTI) AccuSway biomechanics force platform. Participants will be barefoot in an upright stance with arms raised comfortably at their sides, feet abducted, and heels separated. Four posturographic parameters (maximum antero-posterior and medio-lateral displacement, average sway velocity, and 95% confidence ellipse) and two statistical mechanics measures (stabilogram diffusion analysis and detrended fluctuation analysis) will be calculated to quantify postural sway according to our previously published methods.
Time Frame: week 12
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Grip Strength
Description: measure of weakness
Time Frame: week 12
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Gait Speed
Description: Determined based on 4-meter walk at usual speed
Time Frame: week 12
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Strength, Assistance in Walking, Rise From a Chair, Climb Stairs, and Falls (SARC-F) Questionnaire
Description: The SARC-F questionnaire is validated to identify adults with sarcopenia and who are at risk for adverse outcomes and may benefit from a physical function intervention. The scores range from 0 to 10, with 0 to 2 points for each component. A score equal to or greater than 4 is predictive of sarcopenia and poor outcome.
Time Frame: week 12
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Appendicular Lean Muscle Mass/Height
Description: calculated based upon a whole-body DEXA scan performed in the Geriatric Research Unit
Time Frame: week 12
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Community Healthy Activities Model Program for Seniors (CHAMPS) Questionnaire
Description: a brief valid measure that assesses weekly frequency and duration of various physical activities common to older adults to evaluate the efficacy of behavioral interventions to increase levels of physical activity. Caloric expenditure (MET hours/week) will be reported.[8] 'Low activity' will be defined as <6.2 MET-hours/week of activity. Women with MET hr/week between 6.3 and 11.4 will be classified as low-moderate activity. Since only 23% of incontinent women had >11.4 MET hours/week of physical activity, this level will be defined as high activity.
Time Frame: week 12
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Barriers to Physical Activity Questionnaire
Description: Questions regarding attitudes towards physical activity considering UI symptoms and perceived barriers will be assessed. 21-item measure assessing the following barriers to physical activity: 1) lack of time, 2) social influence, 3) lack of energy, 4) lack of willpower, 5) fear of injury, 6) lack of skill, and 7) lack of resources (eg, recreational facilities, exercise equipment). Each domain contains 3 items, with a total score range of 0 to 63 with a higher score indicating a higher amount of perceived barriers.
Time Frame: week 12
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Mobility Assessment Tool-Short Form (MAT-SF) Score
Description: This tool shows self-reported mobility. The score range is 30-80 and a higher score denotes better self-reported mobility.
Time Frame: week 12
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Abdominal Circumference
Description: measure of abdominal circumference will be obtained to determine obesity severity
Time Frame: week 12
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Patient Global Impression of Improvement (PGI)
Description: The PGI is a single-item, 7-point scale used to assess a patient's overall perception of their condition's change after treatment. Originating from the Clinical Global Impression-Improvement (CGI-I) scale used by clinicians, the PGI-I allows patients to rate their progress from "Very Much Improved" to "Very Much Worse," providing a simple, validated, and patient-centered outcome measure for various medical and psychiatric conditions. Scores range from 1 (Very Much Improved) to 7 (Very Much Worse).
Time Frame: week 12
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Patient Satisfaction Question
Description: Participants are asked how satisfied they are with their progress in this program. Score ranges from 1 (Completely) to 3 (Not at all)
Time Frame: week 12
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Estimated Perception of Improvement Question
Description: Participants estimate how much better they are on a scale from 0% (no better) to 100% (completely better).
Time Frame: week 12
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Montreal Cognitive Assessment (MoCA)
Description: MoCA score ranges from 0 to 30 and is used as a screening tool for mild cognitive impairment. A score of 26 or over is considered to be normal.
Time Frame: week 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Collected from baseline through week 12
Arm/Group | Functionally Impaired | Functionally Normal
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/37
Other Adverse Events (participants affected / at risk) | 0/33 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT03057834/Prot_SAP_001.pdf
  • Informed Consent Form (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT03057834/ICF_000.pdf